CLINICAL TRIAL: NCT04065061
Title: Investigation of Erinacine A-enriched Hericium Erinaceus Mycelia for Improvement of Recognition, Vision, and Functional MRI Alterations
Brief Title: Erinacine A-enriched Hericium Erinaceus Mycelia for Improvement of Recognition, Vision, and Functional MRI Alterations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Principal Investigator, David Pei-Cheng Lin, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CS15049
Record Dates: First submitted 2019-08-15; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Supplement; Cognition Disorders in Old Age; Vision; fMRI
Keywords: Erinacine A, supplement, Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Randomized Double Blinded placebo study
Who Masked: Participant, Care Provider, Investigator
Masking Description: to be completed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Erinacine A-enriched Hericium Erinaceus Mycelia dietary supplement from week 0 to week 49.
  Interventions: Dietary Supplement: Erinacine A-enriched Hericium Erinaceus Mycelia
- Placebo (Placebo Comparator): Placebo dietary supplement from week 0 to week 49.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Erinacine A-enriched Hericium Erinaceus Mycelia
  Arms: Experimental
Dietary Supplement: Placebo — Placebo supplement was given to the participants.
  Arms: Placebo

SUMMARY:
This study was designed as randomized double blind placebo study to investigate the efficacy of Erinacine A-enriched Hericium erinaceus mycelia for improvement of recognition, vision, and functional MRI alterations.

DETAILED DESCRIPTION:
Patients were recruited with diagnosis of mild or medium dementia, according to criteria by NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association) as probable or possible Alzheimer's disease. Upon signature of informed consent, they were subject to: (1) Cognitive assessments, including Mini-Mental State Examination(MMSE), Neuropsychiatric Inventory (NPI), Cognitive Abilities Screening Instrument (CASI), and Instrumental Activities of Daily Living (IADL) on weeks 0, 12, 24, and 49, (2) Blood Markers Tests, including DHEAS, Alpha 1-antichymotrypsin, Superoxide Dismutase, and Homocysteine, Apolipoprotein E, Hemoglobin, Calcium, Albumin, and Amyloid Beta on weeks 0, 24, and 49, (3) fMRI Assessments for Super-resolution Track Density Imaging (TDI), and Blood Oxygenation Level-Dependent (BOLD) Signal Mapping, on weeks 0 and 49, (4) Vision Assessments, including Visual Acuity (VA) and Contrast Sensitivity (CS), on weeks 0, 24, and 49. Mann-Whitney U test and Wilcoxon tests were applied to examine the data before and after dietary intake of Erinacine A-enriched Hericium Erinaceus Mycelia after 49 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50 and 90
* Confirmed diagnosis of mild and intermediate Alzheimer's disease based on clinical assessments according to criteria of NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association)

Exclusion Criteria:

* vulnerable to injuries
* loss of self-recognition,
* loss of behavioral capacity
* with critical illness
* with major diseases

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2016-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination(MMSE) | weeks 0,12, 24, and 49
  Assess changes of Mini-Mental State Examination(MMSE) on weeks 0, 12, 24, and 49.
Neuropsychiatric Inventory (NPI) | weeks 0,12, 24, and 49
  Assess changes of Neuropsychiatric Inventory (NPI) on weeks 0, 12, 24, and 49.
Cognitive Abilities Screening Instrument (CASI) | weeks 0,12, 24, and 49
  Assess changes of Cognitive Abilities Screening Instrument (CASI) on weeks 0, 12, 24, and 49.
Instrumental Activities of Daily Living (IADL) | weeks 0,12, 24, and 49
  Assess changes of Instrumental Activities of Daily Living (IADL) on weeks 0, 12, 24, and 49.
Dehydroepiandrosterone sulfate (DHEAS) | weeks 0, 24, and 49
  Assess changes of DHEAS on weeks 0, 24, and 49.
Alpha 1-antichymotrypsin | weeks 0, 24, and 49
  Assess changes of Alpha 1-antichymotrypsinon weeks 0, 24, and 49.
Superoxide Dismutase | weeks 0, 24, and 49
  Assess changes of Superoxide Dismutase on weeks 0, 24, and 49.
Homocysteine | weeks 0, 24, and 49
  Assess changes of Homocysteine on weeks 0, 24, and 49.
Apolipoprotein E | weeks 0, 24, and 49
  Assess changes of Apolipoprotein E on weeks 0, 24, and 49.
Hemoglobin | weeks 0, 24, and 49
  Assess changes of Hemoglobin on weeks 0, 24, and 49.
Calcium | weeks 0, 24, and 49
  Assess changes of Calcium on weeks 0, 24, and 49.
Albumin | weeks 0, 24, and 49
  Assess changes of Albumin on weeks 0, 24, and 49.
Amyloid Beta | weeks 0, 24, and 49
  Assess changes of Amyloid Beta on weeks 0, 24, and 49.
fMRI-Super-resolution Track Density Imaging (TDI) | weeks 0 and 49
  Assess changes of Super-resolution Track Density Imaging (TDI) on weeks 0 and 49.
fMRI-Blood Oxygenation Level-Dependent (BOLD) Signal Mapping | weeks 0 and 49
  Assess changes of Blood Oxygenation Level-Dependent (BOLD) Signal Mapping, on weeks 0 and 49.
Vision Assessments-Visual Acuity (VA) | weeks 0, 24, and 49
  Assess changes of Visual Acuity (VA) on weeks 0, 24, and 49.
Vision Assessments-Contrast Sensitivity (CS) | weeks 0, 24, and 49
  Assess changes of Contrast Sensitivity (CS) on weeks 0, 24, and 49.

CONTACTS AND LOCATIONS:
Overall Officials: David Pei-Cheng Lin, PhD, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li IC, Chang HH, Lin CH, Chen WP, Lu TH, Lee LY, Chen YW, Chen YP, Chen CC, Lin DP. Prevention of Early Alzheimer's Disease by Erinacine A-Enriched Hericium erinaceus Mycelia Pilot Double-Blind Placebo-Controlled Study. Front Aging Neurosci. 2020 Jun 3;12:155. doi: 10.3389/fnagi.2020.00155. eCollection 2020. PMID 32581767